CLINICAL TRIAL: NCT05149287
Title: Early Reduction of Post-opeRative Pain and Inflammation to Expedite Return to Function After KNEE Arthroscopy
Brief Title: PROPER Trial of Pain and Inflammation After Knee Arthroscopy
Acronym: PROPER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding stopped
Sponsor: Austin V Stone (Other)
Responsible Party: Sponsor-Investigator, Austin V Stone, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 63476
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Meniscus Tear; Meniscus Lesion; Cartilage Injury
MeSH Terms: interventions — Ceftriaxone; Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: After providing informed consent, patients undergoing arthroscopy of the knee for meniscal or cartilage injuries will be randomized into one of two groups. At the time of surgery, while the patient is under anesthesia, one group will receive a single intravenous dose of 1 gram of ceftriaxone and the other will receive a single intravenous dose of 1% lidocaine in saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One group will receive an intravenous dose of ceftriaxone and the other will receive an intravenous dose of lidocaine in saline. The syringes will be blinded to ensure that both the investigator administering the injection and the patient will be blinded to the group assignment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): The experimental group will receive a single intravenous dose of 1 g of ceftriaxone immediately postoperative in the operating room.
  Interventions: Drug: Ceftriaxone
- Placebo (Placebo Comparator): The placebo group will receive a single intravenous dose of 1% lidocaine and saline immediately postoperative in the operating room.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ceftriaxone — single intravenous dose of 1 g of ceftriaxone
  Arms: Experimental
Other: Placebo — 1% lidocaine and saline
  Other Names: Lidocaine and Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if ceftriaxone administered postoperatively via intravenous injection reduces postoperative visual analog scale (VAS) pain scores and narcotic consumption in patients undergoing knee arthroscopy for a cartilage or meniscal injury.

DETAILED DESCRIPTION:
Arthroscopic surgery for cartilage and meniscus injuries are some of the most common orthopaedic procedures currently performed. Post-surgical pain is initiated through an inflammatory response to surgery. The pain response leads to sleep disruption and a further increase in pain and additional sleep disruption. Opioid medications are often used after surgery to treat pain despite the side effect profile. These medications also contribute to poor sleep quality and duration. Early pain and narcotic use can be controlled by mitigating the effects of post-surgical inflammation. Ceftriaxone is a readily available antibiotic and may have the desirable anti-inflammatory and analgesic effects, but without the side effects caused by other medications. Since it is highly selective in its inhibition, ceftriaxone is an excellent candidate for reducing immediate post-operative pain and heightened inflammatory response.

By doing this study, the investigators hope to learn about the anti-inflammatory effectiveness of the antibiotic ceftriaxone. Ceftriaxone has been shown to inhibit a key enzyme in the post-operative inflammatory process and has been safely used for treatment of infections for years. The investigators would like to gather information about whether ceftriaxone helps reduce pain and inflammation after surgery. Participation in this research will last about 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study
2. Male or female greater than or equal to 18 years of age and less than 55 years of age
3. Is indicated for knee arthroscopy for cartilage or meniscal procedure
4. Ambulatory and in good general health
5. Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions.
6. Willing to abstain from use of protocol-restricted medications during the study

Exclusion Criteria:

1. Known allergic reactions to cephalosporins
2. Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
3. History of infection in either knee joint
4. Clinical signs and symptoms of active knee infection or crystal disease in either knee within 1 month of Screening
5. Other surgery or arthroscopy of either knee within 6 months of Screening
6. Intraarticular treatment of any joint with any of the following agents within six (6) months of Screening: any corticosteroid preparation or any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection; investigational or marketed).
7. Intraarticular treatment in either knee with hyaluronic acid (investigational or marketed) within 6 months of Screening
8. Parenteral or oral corticosteroids (investigational or marketed) within 3 months of Screening
9. Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening
10. Females who are pregnant or nursing or plan to become pregnant during the study; men whose female partner plans to conceive during the study
11. Radiographic osteoarthritic changes defined as Kellgren-Lawrence grade 2 or greater (as determined by PI from patient's preoperative X-rays)
12. Inability to read and understand English
13. Any prior diagnosis of antibiotic-resistant diarrhea

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Austin V Stone, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
With the participant's approval and as approved by local Institutional Review Boards (IRBs), de-identified biological samples will be stored at the University of Kentucky Orthopedic Biomarker Repository. These samples could be used to research the causes of osteoarthritis after cartilage or meniscus injury, its complications and other conditions for which individuals with cartilage or meniscus injuries are at increased risk, and to improve treatment.
  Before sharing biomarker samples, we will ensure that the participant has given previous consent to the sharing of the information or samples. When we confirm that the previously provided consent is still in effect we will remove identifiers such as (e.g., name, medical record number, or date of birth). We will use a secure electronic log to track information shared without releasing the individual participant's identity.
Supporting Information: Study Protocol
Time Frame: Access to individual participant data will be available 1 year after the final study follow-up has been completed, and will be available until 5 years after the final study follow-up has been completed.
Access Criteria: The researchers requesting access to participant information or samples must complete a questionnaire describing why they need information or samples for their research and how they will use the information or samples. The researchers who receive the information or samples will sign an agreement to use the data responsibly.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (1.5) | 45.5 (9.1) | 43.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Pain Score
Description: The Visual analog scale scores range from 0 to 10 with greater scores indicative of greater pain.
Time Frame: Pre-operative, 2 months post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 3 | 2
units on a scale | -2.67 (1.11) | -2.1 (2.97)

2. Primary Outcome: Change in RU SATED Score
Description: The Regularity, Sleep Quality, Alertness, Timing, Efficiency, Duration scale for sleep (RU SATED) ranges from 0 to 30, with higher scores indicating better sleep health.
Time Frame: Pre-operative, 2 months post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 3 | 2
units on a scale | 1 (0) | -0.5 (2.1)

3. Primary Outcome: Post-operative Narcotic Use
Description: Post-operative narcotic use will be monitored with self-reported medication consumption at the first post-operative visit, which will take place 5-12 days post-operative. The milligrams of morphine equivalent (MME) will be calculated based on patient responses with greater MME indicative of increased postoperative use of narcotic pain medications.
Time Frame: 5-12 days post-operative
Measure: Mean (Standard Deviation); unit: milligrams of morphine equivalent (MME)
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 3 | 2
milligrams of morphine equivalent (MME) | 15 (4.4) | 5.5 (2.1)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT05149287/Prot_SAP_000.pdf